CLINICAL TRIAL: NCT07400055
Title: Evaluation of Medulla Spinalis Edema After CT-Guided Percutaneous Cervical Cordotomy Using Magnetic Resonance Imaging and Its Association With Postprocedural Clinical Outcomes in Patients With Cancer Pain
Brief Title: MRI Evaluation of Spinal Cord Edema After CT-Guided Percutaneous Cordotomy in Cancer Pain Patients
Acronym: CORD-MRI
Status: Not yet recruiting | Type: Observational
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Mesut Bakır, Associate Professor of Anesthesiology and Algology, Mersin University
Other Study IDs: CORD-MRI-2026
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cancer Pain; Intractable Pain; Spinal Cord Edema; Neuropathic Pain
Keywords: Percutaneous Cordotomy; CT-guided Cordotomy; Cervical Cordotomy; Spinal Cord MRI; Radiofrequency Ablation; Postprocedural Complications
MeSH Terms: conditions — Cancer Pain; Pain, Intractable; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Percutaneous Cervical Cordotomy Cohort: Adult patients with cancer-related pain undergoing routine CT-guided percutaneous cervical cordotomy and followed with postoperative MRI and clinical assessments.
  Interventions: Procedure: CT-guided Percutaneous Cervical Cordotomy

INTERVENTIONS:
Procedure: CT-guided Percutaneous Cervical Cordotomy — Routine clinical percutaneous cervical cordotomy performed under CT guidance using radiofrequency ablation at the C1-C2 level for the treatment of intractable cancer pain.

SUMMARY:
This observational study aims to evaluate changes in the spinal cord following CT-guided percutaneous cervical cordotomy performed for the treatment of intractable cancer-related pain. Cordotomy is a routine clinical procedure used to relieve severe pain in selected cancer patients. After the procedure, some patients may develop temporary neurological symptoms that are thought to be related to spinal cord edema.

In this study, magnetic resonance imaging (MRI) will be performed as part of routine clinical follow-up on postoperative day 1 and at 1 month to assess the presence and extent of spinal cord edema. Clinical outcomes, including pain intensity and possible postprocedural symptoms, will be recorded and compared with MRI findings.

The goal of this research is to better understand the relationship between imaging changes in the spinal cord and clinical outcomes after cordotomy, which may help improve patient care and postoperative management in the future.

DETAILED DESCRIPTION:
Percutaneous cervical cordotomy is a well-established palliative procedure used for the management of severe unilateral cancer-related pain that is refractory to medical treatment. The procedure involves CT-guided placement of a radiofrequency electrode at the C1-C2 level to create a lesion in the anterolateral spinothalamic tract, resulting in effective pain relief. Despite its efficacy, transient neurological effects such as dysesthesia, sensory disturbances, and neuropathic pain may occur following the procedure. These clinical findings are believed to be associated with postoperative changes in the spinal cord, including edema.

This prospective observational study is designed to evaluate the presence and extent of medulla spinalis edema following CT-guided percutaneous cervical cordotomy and to investigate its association with clinical outcomes.

A total of 10 to 15 adult patients with cancer-related pain who undergo cordotomy as part of routine clinical care at Mersin University Faculty of Medicine Algology Clinic will be enrolled. Eligible patients will be those aged 18 years or older with an indication for cordotomy.

All procedures will be performed under CT guidance at the C2 level using radiofrequency ablation with standard clinical parameters. No additional interventions will be applied for research purposes.

Clinical assessments will include baseline pain intensity measured using a numeric rating scale (NRS), postoperative pain scores, and evaluation of potential neurological symptoms such as dysesthesia, sensory loss, and other transient complications.

Cervical MRI will be performed as part of routine follow-up on postoperative day 1 and at 1 month. MRI images will be evaluated by a single experienced radiologist who will assess the presence, location, and extent of spinal cord edema and any additional structural changes.

The primary objective is to determine the frequency and characteristics of spinal cord edema following cordotomy as detected by MRI. Secondary objectives include evaluating the relationship between MRI findings and postoperative clinical symptoms as well as changes in pain intensity.

All collected data will be analyzed descriptively and through correlation analyses to explore associations between imaging findings and clinical outcomes.

This study aims to provide a better understanding of postoperative spinal cord changes after cordotomy and their clinical significance, potentially contributing to improved patient selection, monitoring, and management strategies.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years and older

Patients with cancer-related pain refractory to medical treatment

Patients scheduled to undergo CT-guided percutaneous cervical cordotomy as part of routine clinical care

Ability to provide informed consent

Availability for postoperative MRI follow-up on day 1 and at 1 month

Exclusion Criteria:

Patients younger than 18 years

Patients without an indication for percutaneous cervical cordotomy

Inability to undergo MRI (e.g., incompatible implants, severe claustrophobia)

Patients who decline participation or withdraw consent

Incomplete clinical or imaging follow-up data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with intractable cancer-related pain undergoing routine CT-guided percutaneous cervical cordotomy at a tertiary university hospital pain clinic. Participants will be followed prospectively with postoperative MRI and clinical assessments.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Presence and extent of spinal cord edema on cervical MRI after CT-guided percutaneous cordotomy | Postoperative day 1 and 1 month
  Spinal cord edema will be evaluated on cervical MRI by a single radiologist, including presence, location, and longitudinal extent of edema.

SECONDARY OUTCOMES:
Change in pain intensity measured by Numeric Rating Scale (NRS) | Baseline, postoperative day 1, and 1 month
  Pain severity will be assessed using a 0-10 numeric rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mesut Bakır, Principal Investigator — Mersin University Faculty of Medicine, Pain Clinic
Locations (1):
- Mersin University Faculty of Medicine, Department of Algology, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient privacy concerns and institutional data protection policies. Data will be used solely for the purposes of this study and reported in aggregate form.

REFERENCES:
- [Background] Kanpolat Y, Ozdemir M, Al-Beyati E. CT-guided percutaneous cordotomy for intractable pain in what is more than a disease: lung malignancies. Turk Neurosurg. 2013;23(1):81-7. doi: 10.5137/1019-5149.JTN.6980-12.0. PMID 23344872
- [Background] Mercadante S. Intractable pain and cordotomy. BMJ Support Palliat Care. 2020 Sep;10(3):339. doi: 10.1136/bmjspcare-2020-002360. Epub 2020 May 20. No abstract available. PMID 32434924
- [Background] Zomers PJW, Groeneweg G, Baart S, Huygen FJP. Percutaneous Cervical Cordotomy for the Treatment of Cancer Pain: A Prospective Case Series of 52 Patients with a Long-Term Follow-Up. Pain Pract. 2021 Jun;21(5):557-567. doi: 10.1111/papr.12991. Epub 2021 Jan 22. PMID 33350042